CLINICAL TRIAL: NCT05218902
Title: A Prospective/Retrospective Non-Interventional Study of Vidaza® (Azacitidine) in Patients With International Prognostic Scoring System (IPSS) Intermediate-2 and High-risk Myelodysplastic Syndromes, or Chronic Myelomonocytic Leukemia, or Acute Myeloid Leukemia With 20-30% Blasts and Multi-lineage Dysplasia in China
Brief Title: A Study of Azacitidine in Participants With International Prognostic Scoring System (IPSS) Intermediate-2 and High-risk Myelodysplastic Syndromes (MDS), or Chronic Myelomonocytic Leukemia (CMML), or Acute Myeloid Leukemia (AML)
Acronym: DIM Vidaza
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA055-016
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute
Keywords: Myelodysplastic syndromes (MDS); Azacitidine (AZA); Chronic myelomonocytic leukemia (CMML); Acute myeloid leukemia (AML)
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- Retrospectively enrolled cohort: Participants who initiate Azacitidine (AZA) before enrollment
- Prospectively enrolled cohort: Participants who initiate AZA initiation at enrollment

SUMMARY:
The purpose of this study is to assess the safety and effectiveness in the real-world setting among participants who are treated with Azacitidine in accordance with the China Product Label.

DETAILED DESCRIPTION:
This study will have participants both enrolled retrospectively and prospectively for azacitidine (AZA) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of intermediate-2/ high-risk myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMML) or acute myeloid leukemia (AML) with 20-30% bone marrow blasts and multi-lineage dysplasia
* Initiated azacitidine (AZA) treatment per approved China Product Label after April 2017

Exclusion Criteria:

* Contraindicated for the use of AZA according to China Product Label
* Simultaneously participating in a treatment intervention study

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of participants enrolled retrospectively, who initiate azacitidine (AZA) before enrollment and participants enrolled prospectively, who initiate AZA initiation at enrollment.
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 12 Months
Incidence of Serious Adverse Events (SAEs) | Up to 12 Months
Incidence of Adverse Drug Reactions (ADRs) | Up to 12 Months

SECONDARY OUTCOMES:
Best Overall response rate (ORR) defined as the proportion of participants who achieved best response of superior to stable disease | Up to 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Tianjin, Tianjin Municipality, China

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html